CLINICAL TRIAL: NCT06161363
Title: Description of Compliance With Hydroxychloroquine Treatment in Patients With Systemic Lupus Erythematosus in a Hospital Internal Medicine Consultation
Brief Title: Description of Compliance With Hydroxychloroquine Treatment in Patients With Systemic Lupus Erythematosus
Acronym: LES-HYDROXY
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/23/0473
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Lupus Erythematosus

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The Morisky Medication Adherence Scale (MMAS-8): The Morisky Medication Adherence Scale completed by the patients
  Interventions: Other: The Morisky Medication Adherence Scale

INTERVENTIONS:
Other: The Morisky Medication Adherence Scale — The Morisky Medication Adherence Scale will be completed bu the patients

SUMMARY:
The project focuses on non-compliance in patients with systemic lupus erythematosus taking Plaquenil. More than half of patients with chronic illness are not or only poorly compliant with their treatment and lupus is one of them.

The investigators want to use an already validated existing questionnaire in English, the Morisky Medication Adherence Scale 8 (MMAS 8). These results will make it possible, after a multivariate study with reference to the gold standard which is hydroxychloroquinemia, to see which exact questions in the questionnaire can be used in general medicine practices in order to detect less or non-compliant patients as early as possible.

ELIGIBILITY:
Inclusion Criteria:

Age >18 years

* Patient with systemic lupus erythematosus
* Treatment with PLAQUENIL for > 6 months with dosage of hydroxychloroquinemia planned during the consultation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with systemic lupus erythematosus
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-11-16 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Non-compliance with hydroxychloroquine treatment | Day 0
  to describe the non-compliance with hydroxychloroquine treatment with the Morisky Medication Adherence Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Toulouse Hospital, Toulouse, France